CLINICAL TRIAL: NCT00102037
Title: Evaluation of Safety of Activated Recombinant FVII as an Add-On Therapy in Spinal Surgery
Brief Title: Use of Activated Recombinant FVII in Spinal Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: F7SPIN-2180
Record Dates: First submitted 2005-01-19; First posted 2005-01-20 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Acquired Bleeding Disorder; Spinal Fusion
MeSH Terms: interventions — Factor VII

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: eptacog alfa (activated)
  Other Names: activated recombinant human factor VII

SUMMARY:
This trial is conducted in the United States of America (USA). The purpose of this clinical research trial is to understand how safe and effective Recombinant Activated FVII is for reducing bleeding and blood transfusions in patients undergoing spinal fusion surgery.

ELIGIBILITY:
Inclusion Criteria:

* Elective spinal fusion surgery.

Exclusion Criteria:

* History of thrombotic disorders (myocardial infarction, deep vein thrombosis, pulmonary embolism, stroke, disseminated intravascular coagulation or peripheral artery thrombosis)
* Any trauma within the last 3 months leading to hospitalization > 24 hours
* Angina or known coronary artery disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2004-07; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Safety variables | Within 30 days after surgery

SECONDARY OUTCOMES:
Efficacy variables

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (14):
- United States (14):
  - Novo Nordisk Investigational Site, Sacramento, California
  - Novo Nordisk Investigational Site, San Francisco, California
  - Novo Nordisk Investigational Site, Washington D.C., District of Columbia
  - Novo Nordisk Investigational Site, Miami, Florida
  - Novo Nordisk Investigational Site, Atlanta, Georgia
  - Novo Nordisk Investigational Site, Chicago, Illinois
  - Novo Nordisk Investigational Site, Newark, New Jersey
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
  - Novo Nordisk Investigational Site, Pittsburgh, Pennsylvania
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Plano, Texas
  - Novo Nordisk Investigational Site, Charlottesville, Virginia
  - Novo Nordisk Investigational Site, Richmond, Virginia
  - Novo Nordisk Investigational Site, Seattle, Washington

REFERENCES:
- [Result] Sachs B, Delacy D, Green J, Graham RS, Ramsay J, Kreisler N, Kruse P, Khutoryansky N, Hu SS. Recombinant activated factor VII in spinal surgery: a multicenter, randomized, double-blind, placebo-controlled, dose-escalation trial. Spine (Phila Pa 1976). 2007 Oct 1;32(21):2285-93. doi: 10.1097/BRS.0b013e3181557d45. PMID 17906567
- [Result] Hsia CC, Chin-Yee IH, McAlister VC. Use of recombinant activated factor VII in patients without hemophilia: a meta-analysis of randomized control trials. Ann Surg. 2008 Jul;248(1):61-8. doi: 10.1097/SLA.0b013e318176c4ec. PMID 18580208
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com